CLINICAL TRIAL: NCT04601025
Title: The Effect of Different Types of Plant-Based Fiber in a Protein-Containing Meal During Satiety and Hunger States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Hilal Hizli Güldemir, Assist. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CL10840098
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Appetitive Behavior; Satiety
Keywords: appetite; fiber; protein; satiety
MeSH Terms: conditions — Appetitive Behavior | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoghurt (Experimental)
  Interventions: Dietary Supplement: Yoghurt
- Chickpea+Yoghurt (Experimental)
  Interventions: Dietary Supplement: Chickpea+Yoghurt
- Oat+Yoghurt (Experimental)
  Interventions: Dietary Supplement: Oat+Yoghurt

INTERVENTIONS:
Dietary Supplement: Yoghurt — 200 ml plain full-fat yoghurt
  Arms: Yoghurt
Dietary Supplement: Chickpea+Yoghurt — 80 ml plain full-fat yoghurt + 70 gr cooked chickpea
  Arms: Chickpea+Yoghurt
Dietary Supplement: Oat+Yoghurt — 80 ml plain full-fat yoghurt + 100 gr cooked oat
  Arms: Oat+Yoghurt

SUMMARY:
The study was carried out once a week on the same day and for three-week duration, with total of 17 randomly selected participants with ages between 18 and 24 years. The test foods containing different vegetable fiber sources (chickpeas and oats) were given to the participants every week as isocaloric, which have been the control food for a week. The satiety status was evaluated by visual analog scale (VAS) for total of five times as immediately before the test food consumption and at 30, 60, 90 and 120 minutes after consumption. Fasting and postprandial blood glucose levels were measured. A 24-hour retrospective food consumption record was obtained the next day.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-24 years,
* Studying at the university,
* Not smoking,
* Having normal BMI according to the World Health Organization (18.5-24.9 kg / m2),
* Satisfy blood donation criteria,
* Along with not suffering from diabetes,
* Abnormal thyroid problem,
* Gastrointestinal disorder,
* Food allergy or intolerance

Exclusion Criteria:

* Individuals who smoke,
* Follow a special diet program,
* Having eating disorder,
* Vegan or vegetarian,
* Do not consume legumes,
* Having gluten or lactose intolerance,
* Suffering from a chronic disease,
* Pregnant or breastfeeding

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Change of Satiety | 0, 30, 60, 90 and 120 minutes after test food consumption
  Appetite will be examined using visual analog scale (0-10) with five questions: 0 least and 10 greatest
Baseline and postprandial blood glucose concentration | Up to 120. minutes
  Blood glucose concentration before and at the end of 120.minutes after test food intake
Ad libitum lunch intake | End of the 120.minutes
  Quantification of lunch intake after the 120 minutes of test food consumption

SECONDARY OUTCOMES:
Quantification of food intake during the rest of the day | During the 24-hours of experimental day.
  24-hours food consumption record from the end of the ad libitum lunch until the next day 9.00 AM.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)